CLINICAL TRIAL: NCT07348419
Title: Comparison of the Postoperative Analgesic Efficacy of the Quadro-Iliac Plane Block and the Classical Thoracolumbar Interfascial Plane Block in Single-Level Lumbar Disc Surgery: A Prospective Randomized Controlled Trial
Brief Title: Quadro-Iliac vs Thoracolumbar Interfascial Plane Block for Analgesia After Single-Level Lumbar Disc Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OMUKAEK 2025/279
Record Dates: First submitted 2025-12-31; First posted 2026-01-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain; Spinal Stenosis
MeSH Terms: conditions — Acute Pain; Spinal Stenosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Group QİPB (Other): The Quadro-iliac plane block will be performed 30 minutes before lumbar spine surgery
  Interventions: Other: Quadro-iliac plane block
- Active Comparator: Group TLİP (Other): The classical thoracolumbar interfascial plane (TLIP) block will be performed 30 minutes before lumbar spine surgery.
  Interventions: Other: Classical thoracolumbar interfascial plane block

INTERVENTIONS:
Other: Quadro-iliac plane block — Quadro-iliac plane block will be performed under ultrasound guidance before the induction of general anesthesia.
  Arms: Active Comparator: Group QİPB
Other: Classical thoracolumbar interfascial plane block — Classical thoracolumbar interfascial plane block will be performed under ultrasound guidance before the induction of general anesthesia.
  Arms: Active Comparator: Group TLİP

SUMMARY:
The investigators aim to compare the postoperative analgesic efficacy of the classical thoracolumbar interfascial plane block and the Quadro-iliac plane block for postoperative analgesia management after lumbar disc surgery.

DETAILED DESCRIPTION:
Lumbar spinal stenosis can lead to variable signs and symptoms such as back pain, radiating pain to the lower extremities, and reduced walking capacity. Lumbar disc surgery itself causes significant pain due to extensive dissection and muscle retraction during the procedure. A multimodal analgesic approach is preferred for postoperative pain management after lumbar spine surgery. The addition of regional anesthesia techniques can reduce opioid-related side effects and is associated with earlier mobilization, shorter hospital stay, and improved patient satisfaction.

For patients undergoing lumbar disc surgery, the classical thoracolumbar interfascial plane (TLIP) block and the Quadro-iliac plane block (QIPB) provide effective analgesia for postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years,
* Classified as ASA physical status I-III,
* Scheduled to undergo single-level lumbar spinal surgery under general anesthesia
* Who agree to participate in the study by providing written informed consent

Exclusion Criteria:

* History of bleeding diathesis or current anticoagulant therapy
* Known allergy or hypersensitivity to local anesthetics or opioid medications
* Infection at the planned block injection site
* Previous lumbar spine surgery
* History of gabapentinoid or corticosteroid use within the last 3 weeks
* Inability to use a patient-controlled analgesia (PCA) device
* Suspected pregnancy, confirmed pregnancy, or breastfeeding
* Refusal to undergo the procedure or to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected and compared between groups.

SECONDARY OUTCOMES:
Perioperative pain intensity | 24 hours
  Changes in the Numerical Rating Scale (NRS) will be recorded at rest and during movement. The participant's baseline NRS will be recorded, followed by measurements before and after neuraxial positioning and up to 24 hours post-surgery.
  The NRS is a unidimensional measure of pain intensity in adults. It is a segmented numerical version of the Visual Analog Scale (VAS) where the participant selects a whole number (0-10) that best represents the intensity of their pain. The 11-point numerical scale ranges from '0' representing one end of the pain spectrum (e.g. 'no pain') to '10' representing the other end (e.g. 'worst imaginable pain').
Postoperative nausea and vomiting | 24 hours
  Postoperative nausea and vomiting (PONV):
  During follow-up, patients who experience nausea or vomiting will be evaluated using a verbal descriptive PONV scale (0=None, 1=Mild nausea, 2=Moderate nausea, 3=Single episode of vomiting, 4=More than one episode of vomiting).
Quality of recovery 15 scale | 24 hours after surgery
  Postoperative Quality of Recovery 15 in Turkish scale. The QoR-15 (Quality of Recovery-15) questionnaire is a simple and practical tool used to assess postoperative recovery.
  It consists of 15 items, each scored on a numeric scale from 0 to 10, resulting in a total score ranging from 0 to 150.
  Based on the total score, postoperative recovery is categorized as follows:
  136-150: Excellent recovery
  122-135: Good recovery
  90-121: Moderate recovery
  0-89: Poor recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.